CLINICAL TRIAL: NCT03089099
Title: Development of a Prognostic Model for High Volume Metastatic Castration-Resistant Prostate Cancer Patients by Sequentially Analyzing the Expression of Molecular Markers in Circulating Tumor Cells
Brief Title: Expression of Molecular Markers in Circulating Tumor Cells of Metastatic Castration-Resistant Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Bo Dai, Clinical Professor of Department of Urology, Fudan University
Other Study IDs: CTC-mCRPC
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer Metastatic
Keywords: Metastatic Castration-Resistant Prostate Cancer; circulating tumor cells; Prognosis; Liquid biopsy
MeSH Terms: conditions — Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Other: Blood drawing — Blood drawing

SUMMARY:
As prostate cancer progresses into castration-resistant stage from initial hormone-sensitive status, the biological behavior of tumor cells that dissociated from primary lesions changed. Considered a "liquid biopsy," these circulating tumor cells (CTCs) can show how a patient's cancer responded to treatments. The purpose of this study is to determine whether sequentially analyzing the expression of molecular markers in high volume circulating tumor cells in metastatic castration-resistant prostate cancer patients can predict the therapeutic effects and outcomes of these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients
2. 18 yrs and older, and 80 yrs and younger
3. Histologically or cytologically proven prostate adenocarcinoma;
4. Imaging examinations including Emission Computed Tomography (ECT), Positron Emission Tomography (PET) and so on revealed a high-volume disease of patients(A high-volume of disease was defined by the presence of visceral metastases or four or more bone lesions with at least one beyond the vertebral bodies and pelvis)
5. Have been received hormonal therapy and progressed into castration-resistant stage
6. Not yet receiving chemotherapy
7. Patients are willing to participate and can be followed up regularly

Exclusion Criteria:

1. Received the treatment of abiraterone acetate previously
2. Patients received chemotherapy previously
3. Combined with other malignant tumor history (in addition to the skin basal cell carcinoma or other tumors that have been cured more than five years).

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly Diagnosed High Volume Metastatic Castration-Resistant Prostate Cancer.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-04-24 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
overall survival | 2 years
  Overall survival was defined as the period of time from inclusion to death from any cause, or to the last follow up date.

SECONDARY OUTCOMES:
time to prostate specific antigen (PSA) progression | 2 years
  time from inclusion to prostate specific antigen (PSA) progression
time to radiographic progression | 2 years
  time from inclusion to radiographic progression
complete serologic response rate at 3 month and 6 month | 1 year
  prostate specific antigen response rate at 3 month and 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Dai Bo, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No